CLINICAL TRIAL: NCT04977648
Title: A Prospective, Longitudinal Study of the Natural History and Functional Status of Patients With Centronuclear Myopathies
Brief Title: Natural History Study of Patients With Centronuclear Myopathies
Acronym: NatHis-CNM
Status: Withdrawn | Type: Observational
Why Stopped: The first Clinical trial with DYN101 (UNITE-CNM) was early terminated. As a consequence, Dynacure decided to not perform this study.
Sponsor: Dynacure (Industry)
Responsible Party: Sponsor
Other Study IDs: NH-CNM-001
Record Dates: First submitted 2021-05-21; First posted 2021-07-27 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Centronuclear Myopathy
Keywords: Muscular Diseases; Myopathies, Structural, Congenital; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases
MeSH Terms: conditions — Myopathies, Structural, Congenital; Muscular Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and optional biomarker/genetic samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, longitudinal study of the natural disease course intended to recruit approximately 60 patients with centronuclear myopathies (CNM) in Europe and the United States. The duration of the study, including the enrollment period, will be approximately 4 years. Data from the study will be used to characterize the natural disease course of CNM, to identify prognostic variables of the disease and to determine the best outcome measure(s) for the evaluation of future therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinically symptomatic male or female subjects of all ages (newborns included) with a CNM resulting from a documented mutation in the MTM1 or DNM2 gene.
* 2. A written, signed and dated informed consent must be provided to participate in the study. For subjects <18 years, consent of parent(s)/legal guardian(s) is required; informed assent can be obtained from the child according to local regulations.
* 3. Willing and able to comply with all protocol requirements and procedures.

Exclusion Criteria:

* 1. Participation in any other interventional study. Participation in a previous study should be completed at least 4 weeks before the first study visit.
* 2. Currently undergoing or has undergone previous gene therapy or other therapy for CNM.
* 3. Current or past abuse of alcohol or recreational/narcotic drugs (with the exception of caffeine and nicotine), which in the investigator's opinion would compromise the subject's safety and/or compliance with the study procedures.
* 4. Current or relevant history of physical or psychiatric illness, that would make the subject unlikely to comply with the study procedures. (Note: Subjects in a wheelchair are not to be excluded).
* 5. Subject is mentally incapacitated, or parent(s)/legally-authorized representative are legally incapacitated or have limited legal capacity, or have lack of mental capacity to fully understand the protocol requirements and complete all study required procedures.

Min Age: 0 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages (newborns included) with a CNM resulting from mutations in DNM2 or MTM1.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Motor Function Measure (MFM32) for neuromuscular diseases. | Baseline, Up to 36 months
  The MFM32 assessment will be based on subject age. Scoring from 0 (cannot initiate the task) to 3 (performs the task fully).
Change from baseline in the Peak Inspiratory Pressure (PIP). | Baseline, Up to 36 months
  The PIP assessment will be based on subject age and ventilation status. Results will be expressed in cmH2O.
Change from baseline in the in Peak Expiratory Pressure (PEP). | Baseline, Up to 36 months
  The PEP assessment will be based on subject age and ventilation status. Results will be expressed in cmH2O.

SECONDARY OUTCOMES:
Change from baseline in the Pediatric Quality of Life inventory (PedsQL™). | Baseline, Up to 36 months
  The PedsQL™ questionnaire will be completed by the caregivers or by subjects based on subject age.
Change from baseline in the Assessment of Caregiver Experience with Neuromuscular Disease (ACEND). | Baseline, Up to 36 months
  The ACEND questionnaire will be completed by the caregiver for subjects in the study. Scoring from 1 (needs full time assistance) to 6 (needs no assistance).
Change from baseline in the (Pediatric) Eating Assessment Tool-10 ([Pedi]-EAT-10). | Baseline, Up to 36 months
  The (Pedi)-EAT-10 assessment will be completed by the caregiver based on subject age. Scoring from 0 (no problem) to 4 (severe problem).
Change from baseline in the Meaningful Use of Speech Scale (MUSS). | Baseline, Up to 36 months
  The MUSS will be scored by trained site personnel based on the caregiver's or subject's reporting. Scoring from 0 (never) to 4 (always).

IPD SHARING:
Plan to Share IPD: No